CLINICAL TRIAL: NCT06919549
Title: Results of Repair of Triangular Fibrocartilage Complex Tears Using Mini Anchor:
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Khaled Omar, residant doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFCC tear repir
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Triangular Fibrocartilage Complex Tears

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention group (Active Comparator): arthroscopic repair of triangular fibrocartilage complex tears using mini anchor
  Interventions: Procedure: mini anchor

INTERVENTIONS:
Procedure: mini anchor — arthroscopic repair of triangular fibrocartilage complex tears using mini anchor

SUMMARY:
The Triangular fibrocartilage complex (TFCC) is a grouping of ligaments and cartilage in the wrist The TFCC is comprised of six major components: the distal radioulnar ligaments (dorsal and volar), central articular disk, meniscus homolog, ulnar collateral ligament, ECU subsheath, and the ulnolunate (UL)/ulnotriquetral (UT) ligaments.

This is important for wrist motion, stabilization, and overall hand function, including grip strength may progress to persistent pain, instability of the distal radioulnar joint, and arthritis if left untreated..

The TFCC vascularity is supplied by the anterior interosseous and ulnar arteries, although only a quarter of the TFCC is perfused. The limited vascularity of the TFCC, combined with its intricate soft tissue structure and torsional and axial stresses, makes the TFCC prone to frequent injury while maintaining a limited ability to heal.

Injuries like a fall on the outstretched hand or a forced ulnar deviation of the wrist can lead to an acute TFCC tear.

TFCC tears are a common cause of ulnar sided wrist pain and can be caused by chronic degeneration or traumatic injury.

Acute or chronic triangular fibrocartilage complex (TFCC) tears may result in persistent ulnar-sided wrist pain, loss of grip strength, and loss of function for patients.

A combination of clinical history, physical examination, and magnetic resonance imaging (MRI) may be used to diagnose a TFCC lesion, but confirmation of pathology requires an arthroscopic assessment. Arthroscopic assisted repair techniques have revolutionized surgical management Treatment of TFCC using mini anchor arthroscopically providing many benefits.

Functional outcome using Mayo wrist score after arthroscopic repair of triangular fibrocartilage complex tears using mini anchor

ELIGIBILITY:
Inclusion Criteria:

- Peripheral traumatic tears of triangular fibrocartilage complex in both sexes aged from teenagers to sixty.

b. Exclusion criteria:

1. Degenerative tears of triangular fibrocartilage complex. 2. Central- or radial-sided triangular fibrocartilage complex tears. 3. Tears associated with bony injuries.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome using Mayo wrist score | 3 months
  Functional outcome using Mayo wrist score